CLINICAL TRIAL: NCT07003620
Title: Neoadjuvant Immunochemotherapy for Locally Advanced Cervical Cancer: a Prospective, Single-arm, Phase II Clinical Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Lu Huaiwu, Sun Yat-sen Memorial Hospital of Sun Yat-sen University, Guangzhou, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2024-1115-02
Record Dates: First submitted 2025-04-08; First posted 2025-06-04 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Cervical Cancers
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention Arm (Experimental)
  Interventions: Drug: Neoadjuvant immunochemotherapy

INTERVENTIONS:
Drug: Neoadjuvant immunochemotherapy — All patients will receive three cycles of paclitaxel and carboplatin chemotherapy combined with PD-1/PD-L1 inhibitor therapy, followed by open radical hysterectomy and pelvic lymphadenectomy. Postoperative adjuvant therapy (chemotherapy, chemoradiation, or maintenance immunotherapy) will be determined based on pathological assessment. Tumor tissue samples will be collected during treatment for single-cell sequencing analysis.

SUMMARY:
This is a prospective, single-arm, Phase II clinical trial designed to evaluate the efficacy and safety of paclitaxel and carboplatin combined with PD-1/PD-L1 immune checkpoint inhibitors in the treatment of locally advanced cervical cancer. Using single-cell RNA sequencing (scRNA-seq), the study aims to investigate the molecular mechanisms underlying differential treatment responses and optimize personalized therapeutic strategies.

Eligibility Criteria:

Patients with locally advanced cervical cancer (FIGO stages IB3 to IIB) and a primary tumor diameter >4 cm will be enrolled. All patients must have histologically confirmed squamous cell carcinoma, adenosquamous carcinoma, or common adenocarcinoma, an ECOG performance status of 0-1, and no prior treatment.

Outcome Measures:

* Primary endpoint: Objective response rate (ORR), assessing tumor regression.
* Secondary endpoints:Overall survival (OS), progression-free survival (PFS), and incidence of treatment-related adverse events (graded by CTCAE criteria).
* Exploratory endpoint:** Impact of treatment on the tumor microenvironment and gene expression profiles.

Study Intervention:

All patients will receive three cycles of paclitaxel and carboplatin chemotherapy combined with PD-1/PD-L1 inhibitor therapy, followed by open radical hysterectomy and pelvic lymphadenectomy. Postoperative adjuvant therapy (chemotherapy, chemoradiation, or maintenance immunotherapy) will be determined based on pathological assessment. Tumor tissue samples will be collected during treatment for single-cell sequencing analysis.

Sample Size:

The study plans to enroll at least 34 eligible patients. Based on treatment response, patients will be categorized into high-response and low-response groups, with a minimum of 5 cases per group selected for scRNA-seq to ensure robust molecular mechanism analysis. The sample size calculation assumes a historical ORR of 65% and a target ORR of 85%.

ELIGIBILITY:
Inclusion Criteria:

* Patients with locally advanced cervical cancer (FIGO stages IB3 to IIB) and a primary tumor diameter >4 cm will be enrolled.
* All patients must have histologically confirmed squamous cell carcinoma, adenosquamous carcinoma, or common adenocarcinoma.
* ECOG performance status of 0-1.
* no prior treatment.

Exclusion Criteria:

* Patients with a history of other malignant tumors in the past.
* Patients whose clinical data or treatment information is incomplete.
* Patients with severe comorbidities or those who cannot complete follow-up.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-06-29 (Estimated); Primary Completion 2028-10-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 3 months post-treatment

SECONDARY OUTCOMES:
Overall survival | From the initiation of treatment (first dose of neoadjuvant immunochemotherapy) until the date of death from any cause), assessed up to 3 years
progression-free survival | From the initiation of treatment (first dose of neoadjuvant immunochemotherapy) until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years
incidence of treatment-related adverse events | From the initiation of treatment until 30 days after the last dose of neoadjuvant immunochemotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital of Sun Yat-sen University, Guangzhou, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided